CLINICAL TRIAL: NCT03110081
Title: Comparing the Efficacy of Epidural and Quadratus Lumborum Analgesia After Open Nephrectomy Surgery
Acronym: QL Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-1291
Record Dates: First submitted 2017-03-21; First posted 2017-04-12 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Open Nephrectomy Surgery
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quadratus lumborum block (Experimental): Quadratus lumborum (QL) block group will receive a single shot injection of 25 ml 0.25% bupivacaine pre-operatively, followed post-operatively by infusion of ropivacaine 0.2% continuously administered via the QL catheter for at least 48 hours.
  Interventions: Procedure: Quadratus lumborum block
- Epidural analgesia (Active Comparator): Midthoracic catheters will be inserted preoperatively. A bupivacaine 0.1% infusion will be started before the surgical incision, and continuously administered for at least 48 hr at an infusion rate of 5 ml/hr.
  Interventions: Procedure: Epidural analgesia

INTERVENTIONS:
Procedure: Quadratus lumborum block — Quadratus lumborum (QL) block for open partial nephrectomy.
  Arms: Quadratus lumborum block
Procedure: Epidural analgesia — Epidural analgesia for open partial nephrectomy.
  Arms: Epidural analgesia

SUMMARY:
This study aims to assess if Quadratus Lumborum (QL) blocks are non-inferior to epidural analgesia for pain control and opioid consumption through the third postoperative day in patients having open partial nephrectomy. Patients satisfying all inclusion and exclusion criteria will be randomized in a 1:1 ratio to either epidural catheter or QL catheter.

DETAILED DESCRIPTION:
QL blocks with a single shot and catheters infusions may be an alternative to epidural analgesia. However, the relative efficacy, safety, and cost of the two approaches remain unclear.

Epidural analgesia is frequently used as a component of multimodal analgesia for thoracic and abdominal surgery. QL block has been introduced recently as a component of multimodal analgesia for lower thoracic and abdominal surgery. In general, insertion of QL catheter is easier and safer than insertion of epidural catheters. QL catheter management is also less complicated than epidural analgesia (fewer catheter displacements and less hemodynamic compromise) and decreases the level of complexity in postoperative care. Our hypothesis is that the subcostal QL approach with a continuous catheter is non-inferior to epidural analgesia for pain control and opioid consumption in patients having open partial nephrectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

Adults having for open unilateral partial nephrectomy surgery.

Exclusion Criteria:

1. Pregnancy 2. Intolerance or allergy to opioids 3. Previous radical nephrectomy surgery/midline incision 4. Contraindication to epidural analgesia 5. Contraindications to QL block 6. Chronic pain characterized by: i.Opioids use for more than 30 consecutive days within the 3 preoperative months at the dose equal or greater than equivalent of 15 mg of morphine ii.Abdominal pain for more than 6 months, present most days of the week-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | Arrival to post anesthesia care unit until 72 hours after surgery
  Total IV morphine-equivalent doses used, started postoperatively at the time of arrival to post anesthesia care unit until 72 hours after surgery.
Postoperative pain | Arrival to post anesthesia care unit until 72 hours after surgery
  Time-weighted average verbal rating scale for pain until 72 hours after operation as a time-weighted average, based on nursing assessments at four-hour intervals. The verbal rating scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating worst pain imaginable. Time-weighted average pain is defined as the sum of each time interval between two adjacent pain score measurements multiplied by the average of the two corresponding pain scores divided by the time interval between the first and last pain scores.

SECONDARY OUTCOMES:
Patient Global Assessment | Three days after surgery
  Patient global assessment of pain control is measured on an ordinal scale by the patient. Patients can rate their pain control as poor, fair, good, or excellent.
Doses of antiemetic medications administered | Arrival to post anesthesia care unit until the third day after surgery
  Count of the number of antiemetic medications administered.
Duration of postoperative hospitalization | From the date of surgery to hospital discharge, assessed up to 12 months.
  Duration of postoperative hospitalization
Episodes of hypotension | Arrival to post anesthesia care unit until the third day after surgery
  Number of episodes of hypotension during hospital stay, defined by MAP less than 65 mmHg requiring intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Elsharkawy H, Ahuja S, Sessler DI, Maheshwari K, Mao G, Sakr Esa WA, Soliman LM, Ayad S, Khoshknabi D, Khan MZ, Raza S, DeGrande S, Turan A. Subcostal Anterior Quadratus Lumborum Block Versus Epidural Block for Analgesia in Open Nephrectomy: A Randomized Clinical Trial. Anesth Analg. 2021 Apr 1;132(4):1138-1145. doi: 10.1213/ANE.0000000000005382. PMID 33617181